CLINICAL TRIAL: NCT01302522
Title: Mental Practice Impact on Gait and Cortical Organization in SCI
Brief Title: Mental Practice Impact on Gait and Cortical Organization in Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Stephen Page, PhD, University of Cincinnati
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21AT003842-01 (NIH)
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Incomplete Spinal Cord Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Mental practice — All patients in the study will be administered a regimen of locomotor therapy (rehabilitative therapy working on walking). Half of the patients will also be administered a regimen in which they mentally rehearse the exercises that they have just physically performed.
  Other Names: Motor imagery

SUMMARY:
Spinal cord injury (SCI) is a disabling condition that impairs fundamental abilities, such as ambulation, respiration, and toileting. Compromised ambulation is a common, devastating impairment following SCI. Yet, despite the fundamental desire to walk, no conventional rehabilitation regimen reliably improves ambulation after SCI, and many SCI patients do not have reliable transportation access, decreasing community integration and access to needed services, including rehabilitation. Little is also known about the subtle neural events that may predict motor recovery in incomplete SCI patients. This study will test a novel, safe, easy to implement technique that has shown promise in improving gait in incomplete SCI patients. The investigators expect that this study will confirm the efficacy of this technique, by showing that it increases the speed and efficiency of walking. This outcome is expected to produce a therapy that improves outcomes and health, and reduces care costs, for community dwelling patients with incomplete SCI.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old;
* incomplete SCI (ASIA Grade C or D), experienced > 1 year prior to enrollment;
* motor grade of > 1 < 3 in the quads, hamstrings, and hip flexors, and ability to ambulate with at least a maximal assist;
* range of motion in the lower limbs within functional limits;
* motor function in at least half of ASIA key lower extremity muscles with strength < or > 3/5;
* able to ambulate at least 10 meters with 1 person assistance and/or assistive device;
* medically stable (ie, no bladder infection; decubiti); (8) stable dosage of antispasticity medications for duration of study

Exclusion Criteria:

* excessive spasticity in the lower limbs as measured by a score of > 3 on the Modified Ashworth Spasticity Scale;
* excessive pain in the lower limbs as measured by a score of > 5 on a Visual Analog Scale or > 8/10 with a clarified scaled picture graph;
* moderate to severe osteoporosis, as indicated by the patient's physician;
* heterotropic ossification, as indicated by the patient's physician;
* psychological conditions that would contraindicate participation in the program and no abnormalities of attention, with minimum cognitive capacity present sufficient to participate in MP;
* fracture or fracture history in the lower limbs (individuals with a remote history of fractures may be included at discretion of the study physical therapists at each site);
* enrolled in any form of rehabilitation;
* for subjects to be administered fMRI, implant containing electrical circuitry, generating electrical signals, or having moving metal parts, metal pins or plates above the waist, orthodontic braces, or other positives on a standard checklist of MRI exclusion criteria used by the Radiology Department;
* pregnant;
* DSM-IV Major Depressive Episode symptom criteria of > 5/9 as exclusion threshold instead of CESD;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Gait velocity: The investigators are measuring the speed that people walk. | 1-3 weeks before intervention; 1 week after intervention; 3 months after intervention